CLINICAL TRIAL: NCT01842932
Title: Usefulness Of Flospan As A Premedication For Colonoscopy : A Randomized Double Blind Controlled Trial
Brief Title: Usefulness Of Flospan As A Premedication For Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sun Gyo Lim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AJIRB-MED-CT4-09-257
Record Dates: First submitted 2013-04-14; First posted 2013-04-30 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Anticholinergics
MeSH Terms: interventions — Phloroglucinol; cimetropium; Cholinergic Antagonists; Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phloroglucin & Placebo (Experimental): Phloroglucin 20ml before examination & Placebo 1ml before examination
  Interventions: Drug: Phloroglucin; Procedure: Colonoscopy; Drug: Placebo
- Cimetropium bromide & Placebo (Experimental): Cimetropium bromide 1ml before examination & Placebo 20ml before examination
  Interventions: Drug: Cimetropium bromide; Procedure: Colonoscopy; Drug: Placebo

INTERVENTIONS:
Drug: Phloroglucin — Premedication of colonoscopy
  Other Names: Flospan
  Arms: Phloroglucin & Placebo
Drug: Cimetropium bromide — Premedication of colonoscopy
  Other Names: Anticholinergics; Algiron
  Arms: Cimetropium bromide & Placebo
Procedure: Colonoscopy — Diagnostic examination of colon
  Other Names: Diagnostic examination of colon
Drug: Placebo — Placebo for double-blind study These are harmless to the human body, and are composed of saline solution without drug efficacy.

SUMMARY:
Usefulness of Flospan as a premedication for colonoscopy: A randomized double-blind controlled trial

DETAILED DESCRIPTION:
Cimetropium bromide is premedication of colonoscopy. However, it is contraindication for some diseases; benign prostatic hyperplasia(BPH) or other obstructive uropathy, intestinal obstruction, pyloric stenosis, glaucoma, myasthenia gravis, megacolon, paralytic ileus. In this cases, Flospan (phloroglucin) is effective alternative drug. So our research was to compare the effects of these two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Recipient endoscopic diagnostic purposes.

Exclusion Criteria:

* If you currently pregnant, or of childbearing potential
* Previous abdominal surgery or bowel resection.
* If under 18 years of age
* If the last two days, the administration of anticholinergic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Non inferiority of phloroglucin to cimetropium bromide | Up to ten months
  Comparing the two groups of time of examination, frequency of peristalsis, Scoring for the experimenter and the subject of the inspection feedback, double-blind setting.

SECONDARY OUTCOMES:
Total diagnostic colonoscopy exam time | 1 year
Evaluation of practitioners | 1 year
  Colonic motility and test difficulty
Evaluation of subjects | 1 year
  The degree of discomfort after test
Peristalsis time of transverse colon | 1 year
  Total peristalsis time of transverse colon for two minutes
Total dose and times of sedatives for pain control | 1 year
  Total dose and times of sedatives (midazolam, propofol) for pain control
Time of cecal intubation | 1 year
  Total time of colonoscope intubation from anus to cecum

OTHER OUTCOMES:
Bowel cleansing status | 1 year
Heart rate, respiratory rate, oxygen saturation, blood pressure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kee Myung Lee, M.D., Ph.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea